CLINICAL TRIAL: NCT01432912
Title: Pilot Study Evaluating the Influence of Physician Education Regarding the 5A's Smoking Cessation Counselling Strategy, as Evaluated by Patient Interpretation of the Strategy Principles
Brief Title: Study Evaluating the Effect of Physician Education on Smoking Cessation Counselling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assuta Hospital Systems (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: Maccabi-14/2011
Record Dates: First submitted 2011-09-11; First posted 2011-09-13 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2011-09

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients (No Intervention)
  Interventions: Behavioral: Physician Educational Seminar

INTERVENTIONS:
Behavioral: Physician Educational Seminar — Participating Physicians will attend an hour long seminar on smoking cessation counselling.

SUMMARY:
The purpose of the study is to see if a short seminar educating physicians about smoking cessation counselling will effectively improve their smoking counselling cessation practices.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18yrs and over that visit the participating physicians and agree to compete the study questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2011-09; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Patient assessment questionnaires | Within a month after the seminar.

CONTACTS AND LOCATIONS:
Locations (1):
- Maccabi Healthcare Services, Modiin, Israel